CLINICAL TRIAL: NCT03071627
Title: Interpretation of Health News Items Reporting Results of Pre-clinical Studies With or Without Spin: A Randomized Controlled Trial Among French-speaking Population
Brief Title: Interpretation of Health News Items Reporting Results of Pre-clinical Studies With or Without Spin By French-speaking Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Principal Investigator, Isabelle BOUTRON, Professor, Assistance Publique - Hôpitaux de Paris
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ISB-002
Record Dates: First submitted 2017-02-13; First posted 2017-03-07 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: The Study Focus on no Specific Condition
Keywords: Spin; Misleading reporting; Misleading interpretation; Misleading extrapolation; Animal studies; Cell culture studies; Pre-clinical studies
MeSH Terms: interventions — spindlin

STUDY DESIGN:
Intervention Model Description: Two arms, parallel group, randomized controlled trial
Who Masked: Participant
Masking Description: Participants will be blinded to the study hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- News with Spin (Active Comparator): News items reporting results of animal studies with spin.
  Interventions: Other: New items with spin
- News without spin (Experimental): News items reporting results of animal studies without spin.
  Interventions: Other: New items without spin

INTERVENTIONS:
Other: New items with spin — Interpretation of news items with spin
  Arms: News with Spin
Other: New items without spin — Interpretation of news items without spin
  Arms: News without spin

SUMMARY:
The main objective of this study is to compare the interpretation of health news items reporting results of pre-clinical studies with or without spin (i.e., distortion of research results). The news items which reported those studies evaluating the treatment effect either in cell culture studies or animal studies, have high number of spin in the headline and text and received high online public attention will be selected. Spin will be deleted and will rewrite the news items without spin. This sample of news items reporting results of pre-clinical studies with and without spin will be interpreted by French-speaking population.

DETAILED DESCRIPTION:
Health news is an important way to communicate updated medical research to the public. News items reporting the results of medical research attract a large audience. However, the quality of reporting in health news is questionable. The merits of a wide range of treatments and tests are overplayed and harms are underplayed. Several studies have shown the presence of spin (i.e., distorted presentation of study results) in health news. Distorted facts can be misleading and can affect the behaviour of physicians, healthcare providers and patients. However, little research has assessed whether spin can affect readers' interpretation of health news items.

Objective: To compare the interpretation of health news items reported with or without spin. News items reporting pre-clinical studies evaluating the effect of a pharmacological treatment that received high online public attention will be focused. "Spin" is defined as a misrepresentation of study results whatever the motive (intentionally or unintentionally) to highlight that the beneficial effect of the intervention in terms of efficacy and safety is greater than that shown by the results.

Hypothesis: The hypothesis of this study is that the spin can influence the reader's interpretation of health news items reporting results of pre-clinical studies.

Design: A randomized controlled trial

1. Interventions: Health news items reporting results of pre-clinical studies with and without spin will be compared. A sample of health news items reporting the results of pre-clinical studies evaluating the effect of pharmacologic treatment and containing spin in the headline and text will be selected. Spin will be deleted in the selected news items and will be rewritten the news without spin.
2. Participants: The participants will include French-speaking healthy population from Nutrinet santé.
3. Sample size: For this RCT, the sample size will be 300 participants.
4. Main outcome measures: The primary outcome will be participants' interpretation of the benefit of treatment after reading the news (What do you think is the probability that treatment X would be beneficial to patients? (scale, 0 [very unlikely] to 10 [very likely]).
5. Expected results: This study will evaluate the impact of spin on the interpretation of news items reporting results of pre-clinical studies by French-speaking population.
6. This study is approved by ethics review regulations by INSERM (CEEI-IRB): IRB00003888

ELIGIBILITY:
Inclusion Criteria:

* Native French speakers who can read the news

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Perception of beneficial effect of the treatment X. We ask participants, What do you think is the probability that treatment X would be beneficial to patients? | As the intervention is assigned (reading the news item) i.e., 1-2 hours
  With the choices of answers on a 10 points Likert scale, (scale, 0 [very unlikely] to 10 [very likely])

SECONDARY OUTCOMES:
Perception of efficacy, safety, availability and clinical utility in existing clinical practice for the treatment X. We will ask the participants: What do you think is the size of the potential benefit for patients? | As the intervention is assigned (reading the news item) i.e., 1-2 hours
  With the choice of answers on a 5 points scale, (scale, [none, small, moderate or large]) -- analysis none, small vs moderate, large
How safe do you think that treatment X would be for patients? | As the intervention is assigned (reading the news item) i.e., 1-2 hours
  With the choices of answers on a 10 points Likert scale, (scale, 0 [very unsafe] to 10 [very safe])
Do you think this treatment should be offered to patients in the short term? | As the intervention is assigned (reading the news item) i.e., 1-2 hours
  With the choices of answers on a 10 points Likert scale, (scale, 0 [absolutely no] to 10 [absolutely yes])
Do you think this treatment will make a difference in the existing clinical practice? | As the intervention is assigned (reading the news item) i.e., 1-2 hours
  With the choices of answers on a 10 points Likert scale, (scale, 0 [absolutely no] to 10 [absolutely yes])

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.etude-nutrinet-sante.fr